CLINICAL TRIAL: NCT00353522
Title: A Phase II, Double-Blind, Randomized, Placebo-controlled, Parallel Group Study, Evaluating the Efficacy and Safety of RO4607381 Over a 24-week Period in Patients With CHD or a CHD Risk Equivalent
Brief Title: A Study of RO4607381 in Patients With Coronary Heart Disease (CHD) or a CHD Risk Equivalent.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC19453
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dalcetrapib (Experimental): Dalcetrapib 900mg po daily for 24 weeks
  Interventions: Drug: dalcetrapib
- Placebo (Placebo Comparator): Placebo po daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — po daily for 24 weeks
  Arms: Placebo
Drug: dalcetrapib — 900mg po daily for 24 weeks
  Arms: Dalcetrapib

SUMMARY:
This 2 arm study will investigate the efficacy and safety of RO4607381 in patients with coronary heart disease, or CHD risk equivalent. After a pre-randomization phase of 5-12 weeks, patients will be randomized to receive either RO4607381 (900mg po) or placebo po daily for 24 weeks, with concomitant atorvastatin 10-80mg daily, and changes in cholesterol level and lipoprotein metabolism will be measured. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* CHD or CHD risk equivalent;
* body weight <125kg at visit 1.

Exclusion Criteria:

* recent (within 3 weeks of screening) clinically significant coronary events;
* history of statin-associated myopathy, or intolerance to statin;
* history of malignancy (except for curatively treated basal cell or squamous cell cancer of the skin) during the 3 years prior to screening;
* exposure to RO4607381 in past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (9):
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Bethesda, Maryland
  - Minneapolis, Minnesota
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Salt Lake City, Utah
- Germany (7):
  - Berlin
  - Bochum
  - Dortmund
  - Erlangen
  - Freiburg im Breisgau
  - Hamburg
  - München

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalcetrapib | Placebo
Started | 89 | 46
Completed | 74 | 37
Not Completed | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib | Placebo | Total
Number analyzed (Participants) | 89 | 46 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (7.76) | 60.2 (7.50) | 60.9 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 8 | 29
  Male | 68 | 38 | 106

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in HDL-C
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 89 | 45
mg/dL | 12.76 (1.17) | 0.50 (1.49)

2. Secondary Outcome: Percent Change From Baseline in Cholesterol Ester Transfer Protein (CETP) Mass
Time Frame: Baseline and Weeks 24
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 52 | 25
Percent change | 86.45 (6.30) | -4.93 (8.32)

3. Secondary Outcome: Change in Mesenteric Lymph Nodes
Time Frame: Baseline and 48 Weeks
Measure: Number; unit: Number of Nodes
Units Other Than Participants: Number of Mesenteric Lymph Nodes
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 52 | 25
Number analyzed (Number of Mesenteric Lymph Nodes) | 84 | 41
Number of Nodes
  Number Increased in Volume | 4 | 11
  Number Decreased in Volume | 6 | 18

4. Secondary Outcome: Change From Baseline in Total Cholesterol (TC), Triglycerides (TG), HDL-C, LDL-C, Apolipoproteins A1 (ApoA1), Apolipoproteins B (ApoB)
Time Frame: Baseline and 48 Weeks
Measure: Least Squares Mean (Standard Error); unit: Percent change in mg/dL
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 52 | 25
Percent change in mg/dL
  Total Cholesterol | 10.17 (3.20) | 2.67 (4.22)
  Triglycerides | 0.94 (8.76) | 4.11 (11.63)
  HDL-C | 33.76 (4.43) | 3.69 (5.81)
  LDL-C | 4.75 (4.45) | 2.97 (5.87)
  ApoA1 | 16.43 (2.54) | 8.15 (3.30)
  ApoB | 4.98 (3.83) | 2.48 (5.00)

5. Secondary Outcome: Change From Baseline in Cholesterol Ester Transfer Protein (CETP) Activity
Time Frame: Baseline and 48 Weeks
Measure: Least Squares Mean (Standard Error); unit: percent change in pMOL/mcL/hr
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 52 | 25
percent change in pMOL/mcL/hr | -56.5 (5.09) | -5.69 (6.67)

6. Primary Outcome: Percent Change From Baseline in HDL-C
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Dalcetrapib | Placebo
Number analyzed (Participants) | 89 | 45
Percent Change | 33.40 (2.86) | 3.59 (3.64)

ADVERSE EVENTS:
Arm/Group | Dalcetrapib | Placebo
Serious Adverse Events (participants affected / at risk) | 11/89 | 6/46
Other Adverse Events (participants affected / at risk) | 0/89 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalcetrapib (N=89) | Placebo (N=46)
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OsteoArthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Nerocysterosis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No